CLINICAL TRIAL: NCT00224523
Title: A Randomized, Open Label, Active Controlled (Mometasone Furoate Aqueous Nasal Spray [Nasonex®] 200mcg QD), Parallel Group, Multi-Center, 52-Week Study to Assess the Long Term Safety of GW685698X Aqueous Nasal Spray 100mcg QD Via Nasal Biopsy in Subjects 18 Years of Age With Perennial Allergic Rhinitis (PAR)
Brief Title: Long Term Safety Of GW685698X Via Nasal Biopsy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FFR104503
Record Dates: First submitted 2005-08-26; First posted 2005-09-23 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Rhinitis, Allergic, Perennial
Keywords: perennial allergic rhinitis; nasal biopsy; GW685698X
MeSH Terms: conditions — Rhinitis, Allergic, Perennial | interventions — Mometasone Furoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: GW685698X; Drug: mometasone furoate

INTERVENTIONS:
Drug: GW685698X
Drug: mometasone furoate
  Other Names: GW685698X

SUMMARY:
Long term safety (52 weeks) of GW685698X on the nasal mucosa via nasal biopsy with an active control group (Nasonex®) and a healthy volunteers control group in subjects 18 years old with perennial allergic rhinitis . Allergic rhinitis is an inflammatory disorder of the upper airway that occurs following allergen exposure. Perennial allergic rhinitis is triggered by house dust mites, animal dander, etc., possibly causing symptoms year-round including nasal congestion, rhinorrhea and/or nasal itching.

DETAILED DESCRIPTION:
A Randomized, Open Label, Active Controlled (Mometasone Furoate Aqueous Nasal Spray [Nasonex®] 200mcg QD), Parallel Group, Multi-Center, 52-Week Study to Assess the Long Term Safety of GW685698X Aqueous Nasal Spray 100mcg QD via Nasal Biopsy in Subjects >18 Years of Age with Perennial Allergic Rhinitis (PAR)

ELIGIBILITY:
Inclusion criteria:

* History of perennial allergic rhinitis of 2 years, with a documented positive allergen test to an appropriate allergen.
* Female patients of child-bearing potential must be willing to consistently and correctly use an acceptable method of birth control.

Exclusion criteria:

* Patients who require certain medications for their allergy.
* Patients with serious medical problems.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2005-09; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Quantitative and qualitative differences in the morphology and cytology of the nasal mucosa after 1 year of treatment.

SECONDARY OUTCOMES:
No Secondary Outcome Measures

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- GSK Investigational Site, Leuven, Belgium
- Netherlands (3):
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Nijmegen
  - GSK Investigational Site, The Hague

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Fokkens W, Hellings P, Blom H, Jansen A, van Drunen K, Clements D, Wu W, Caldwell M, Philpot E. A comparison of the effects of fluticasone furoate and mometasone furoate nasal sprays on the nasal mucosa. Ann Allergy Asthma Immunol 2008; 100(1) (Supplement 1):A12 (abstract)
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: FFR104503 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: FFR104503 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: FFR104503 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: FFR104503 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: FFR104503 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: FFR104503 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: FFR104503 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register